CLINICAL TRIAL: NCT00265824
Title: Phase III Study of an Optimized Chemotherapy Followed by Maintenance With Bevacizumab Strategy With or Without Erlotinib in Unresectable Metastatic Colorectal Cancer. DREAM OPTIMOX 3. C04-2
Brief Title: Optimized Chemotherapy Followed by Maintenance With Bevacizumab With or Without Erlotinib in Treating Patients With Metastatic Colorectal Cancer That Cannot be Removed by Surgery (DREAM)
Acronym: DREAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000453861; GERCOR-C04-2; EU-20565; GERCOR-OPTIMOX3; GERCOR-DREAM- C04-2
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2014-03

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bevacizumab alone (Active Comparator)
  Interventions: Drug: bevacizumab
- Bevacizumab + erlotinib (Experimental)
  Interventions: Drug: bevacizumab, erlotinib

INTERVENTIONS:
Drug: bevacizumab — bevacizumab 7.5mg/kg every 3 weeks until disease progression or limiting toxicity
  Arms: bevacizumab alone
Drug: bevacizumab, erlotinib — bevacizumab 7.5mg/kg and oral erlotinib 150 mg/day continuously Cycles every 3 weeks until disease progression or limiting toxicity
  Arms: Bevacizumab + erlotinib

SUMMARY:
PURPOSE: This randomized phase III trial is studying maintenance therapy with bevacizumab alone after an induction therapy combining bevacizumab+chemotherapy to see how well they work compared to maintenance therapy with bevacizumab+erlotinib alone after an induction therapy combining bevacizumab+chemotherapy in treating patients with metastatic colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare Progression-free survival during maintenance period ("Maintenance PFS")in patients with unresectable metastatic colorectal cancer.

Secondary

* Compare the duration of disease control and overall survival of patients treated with these regimens.
* Compare the tolerability of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare the occurrence of secondary surgery in patients treated with these regimens.
* Compare the chemotherapy-free intervals and response rates in patients treated with these regimens.

INDUCTION THERAPY

Bevacizumab IV over 30-90 minutes on day 1, combined with either:

* modified FOLFOX7 (IV : oxaliplatin, folinic acid, fluorouracil),
* XELOX2 (IV : oxaliplatin, oral capecitabine day 1 to 8),
* FOLFIRI (IV : irinotecan, folinic acid, fluorouracil).

Treatment repeats every 2 weeks.

RANDOMIZATION Patients with stable or responding disease then receive maintenance therapy with bevacizumab alone or bevacizumab+erlotinib

MAINTENANCE THERAPY

* Arm A : bevacizumab alone : bevacizumab IV over 30-90 minutes on day 1
* Arm B : bevacizumab+erlotinib : bevacizumab IV over 30-90 minutes on day 1 and oral erlotinib once daily on days 1-21.

In both arms, treatment with bevacizumab +/- erlotinib repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

ACCRUAL: A total of 700 patients will be accrued for this study.

ELIGIBILITY:
MAIN ELIGIBILITY CRITERIA

* Histologically proven metastatic adenocarcinoma of colon or rectum
* Documented inoperable disease (i.e., not suitable for complete carcinological surgical resection)
* Measurable lesion as assessed by CT scan or MRI in at least one dimension (longest diameter to be recorded) ≥ 20 mm with conventional CT scan or ≥ 10 mm with spiral CT scan
* No previous therapy for metastatic disease
* No history or evidence upon physical examination of CNS disease (e.g., non-irradiated CNS metastasis, seizure not controlled with standard medical therapy, or history of stroke) unless adequately treated
* No exclusive bone metastasis
* ECOG performance status 0-2
* WBC ≥ 1,500/mm^3
* Platelets ≥ 100,000/mm^3
* Hemoglobin > 9 g/dL (may be transfused to maintain or exceed this level)
* Proteinuria < 2+ by dipstick OR ≤ 1 g of protein on 24-hr urine collection
* Bilirubin < 1.5 times ULN
* Alkaline phosphatase < 3 times ULN
* No peripheral sensory neuropathy
* Negative pregnancy test
* Fertile patients must use effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly, or surgically sterilization)
* No peripheral neuropathy ≥ grade 1
* No clinically significant (i.e. active) cardiovascular disease
* No evidence of bleeding diathesis or coagulopathy
* No serious, non-healing wound, ulcer, or bone fracture
* No significant ophthalmologic abnormality
* More than 28 days since prior major surgical procedure or open biopsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2005-05; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival during maintenance therapy | Tumor evaluation every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Aimery de Gramont, MD, Study Chair — Hopital Saint Antoine; Christophe Tournigand, MD, Study Chair — Hopital Henri Mondor
Locations (47):
- Austria (4):
  - LKH Leoben, Leoben
  - LKH Steyr, Steyr
  - AKH Universitätsklinik für Innere Medizin I, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Canada (6):
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Cité de la Santé de Laval, Laval, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM Hôpital Notre-Dame, Montreal, Quebec
  - Mc Gill University Hospital, Montreal, Quebec
  - Hôpital Charles LeMoyne, Montreal, Quebec
- France (37):
  - Centre Hospitalier, Antibes
  - Centre Hospitalier, Auxerre
  - Centre Hospitalier, Beauvais
  - Hôpital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre Hospitalier, Briey
  - Hôpital Pasteur, Colmar
  - Centre Hospitalier, Dax
  - Hopital Drevon, Dijon
  - CHD les oudairies, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - Hopital Robert Boulin, Libourne
  - CHU Dupuytren, Limoges
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Clinique de la sauvegarde, Lyon
  - hôpital Ambroise Paré, Marseille
  - Institu Paoli Calmette, Marseille
  - Centre Hospitalier, Meaux
  - Clinique Claude BERNARD, Metz
  - Centre hospitalier Layné, Mont-de-Marsan
  - Centre Hospitalier Intercommunal Le Raincy - Montfermeil, Montfermeil
  - centre oncologie de Gentilly, Nancy
  - Centre Catherine de Sienne, Nantes
  - Institut Curie, Paris
  - Groupe Hospitalier les Diaconnesses, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Saint Joseph, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - centre Catalan oncologie, Perpignan
  - Clinique Armoricaine, Saint-Brieuc
  - Centre Hospitalier, Semur-en-Auxois
  - C.H. Senlis, Senlis
  - Hopital Foch, Suresnes
  - Clinique Générale, Valence

REFERENCES:
- [Derived] Tournigand C, Chibaudel B, Samson B, Scheithauer W, Vernerey D, Mesange P, Lledo G, Viret F, Ramee JF, Tubiana-Mathieu N, Dauba J, Dupuis O, Rinaldi Y, Mabro M, Aucoin N, Latreille J, Bonnetain F, Louvet C, Larsen AK, Andre T, de Gramont A. Bevacizumab with or without erlotinib as maintenance therapy in patients with metastatic colorectal cancer (GERCOR DREAM; OPTIMOX3): a randomised, open-label, phase 3 trial. Lancet Oncol. 2015 Nov;16(15):1493-1505. doi: 10.1016/S1470-2045(15)00216-8. Epub 2015 Oct 22. PMID 26474518